CLINICAL TRIAL: NCT00944177
Title: Study to Evaluate the Bioequivalence of a Test Tablet Formulation of Metformin HCl (1000 mg), Compared to an Equivalent Dose of a Commercially Available Reference Drug Product (Glucophage®, Bristol-Myers Squibb Company) in Fasted, Healthy, Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Torrent Pharmaceuticals Limited (Industry)
Other Study IDs: 40483
Record Dates: First submitted 2009-07-21; First posted 2009-07-23 (Estimated); Last update posted 2009-07-23 (Estimated); Status verified 2009-07

CONDITIONS: Healthy
MeSH Terms: interventions — Metformin

INTERVENTIONS:
Drug: Metformin HCl

SUMMARY:
* Objective:

  * A Randomized, Two-Way Crossover, Single-Dose, Open-Label Study to Evaluate the Bioequivalence of a Test Tablet Formulation of Metformin HCl (1000 mg), Compared to an Equivalent Dose of a Commercially Available Reference Drug Product (Glucophage®, Bristol-Myers Squibb Company) in Fasted, Healthy, Adult Subjects.
* Study Design:

  * Randomized,single-dose,2-way crossover.

ELIGIBILITY:
Inclusion Criteria:

* Subject is at least 18 years old.
* Subject had no clinically significant abnormal lab values at the screening evaluation.
* Subject's drugs of abuse, Hepatitis B, Hepatitis C, and HIV screenings were negative or non-relative.
* Acceptable screening of ECG.
* Female subject's pregnancy test at screening is negative.
* Subject had no evidence of underlying disease at the pre-entry physical examination.
* Subject has given written consent to participate.
* Female subject has not received any injectable or implantable contraceptive for a period of six months preceding this study.
* Agreed to undergo at least a 14-day pre-dose washout.
* Beginning two weeks prior to dosing and throughout the study, female subject of childbearing potential agrees to utilize one of the following methods of contraception:

  1. Condom and topical spermicide
  2. Condom and diaphragm
  3. Intra-uterine device (I.U.D)
  4. Complete abstinence.
* Agree to abstain from consuming caffeine or alcohol for at least 48 hours. prior to study and throughout the blood collection periods.

Exclusion Criteria:

* History of treatment for alcoholism, substance abuse, or drug abuse with in the past 24 months.
* History of malignancy, stroke, diabetes, cardiac, renal or liver disease, or other serious illness.
* History of GRD, malabsorption syndrome, colon cancer, or chronic colitis, including Crohn's disease.
* History of treatment for asthma, hypoxemia, dehydration, sepsis, metabolic acidosis and congestive heart failure.
* Subject is pregnant or lactating.
* History of drug hyper sensitivity.
* Subject was treated with any investigational drug during the four weeks prior to initial dosing for the study.
* Subject smokes more then 15 cigarettes per day or uses tobacco products or currently uses nicotine products.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Gateway Medical Research, Inc., Saint Charles, Missouri, United States